CLINICAL TRIAL: NCT07344220
Title: Metastatic Non-Familial Adenocarcinoma Maintenance Therapy With DZ-002: Heptamine Carboxymethine Dye Conjugate
Acronym: DZ-002-201
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Collaborators: Da Zen Theranostics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 132-25-CA; DZ-002-201 (Other: Hoag Memorial Hospital Presbyterian)
Record Dates: First submitted 2025-11-12; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Pancreatic Cancer
Keywords: Dose Escalation Phase; Dose Maintenance Phase; Recommended Phase 2 Dose; RP2D
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The first 3-6 participants taking part in this study will receive the lowest dose of study drug 5mg/kg. If the study drug does not cause unmanageable side effects at the 5mg/kg dose level, the next group of 3-6 participants will receive a higher dose of study drug 6mg/kg. If the study drug does not cause unmanageable side effects at the 6mg/kg dose level, the next group of 3-6 participants will receive the highest dose of study drug 7mg/kg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Phase (Experimental): First 9-18 patients will be enrolled on the dose escalation portion. Starting dose: 3-6 study participants 5 mg/kg iv weekly Second dose: 3-6 study participants 6 mg/kg iv weekly Final dose: 3-6 study participants 7 mg/kg iv weekly
  Interventions: Drug: DZ-002 - 5 mg/kg, 6 mg/kg, or 7 mg/kg
- Maintenance Phase (Experimental): Additional 30 patients will be enrolled and receive the RP2D from the dose escalation phase. All patients will receive the iv weekly selected RP2Dose from dose escalation portion.
  Interventions: Drug: DZ-002 - 5 mg/kg, 6 mg/kg, or 7 mg/kg

INTERVENTIONS:
Drug: DZ-002 - 5 mg/kg, 6 mg/kg, or 7 mg/kg — 5 mg/kg, 6 mg/kg, or 7 mg/kg DZ-002 administered by IV over a 4-hour period, on Days 1, 8, 15, and 22 of a 4-week period, or cycle.

SUMMARY:
The goal of this clinical trial is to learn if drug DZ-002 works to treat adults with metastatic pancreatic adenocarcinoma. It will also learn about the safety of drug DZ-002. The main questions it aims to answer are:

* To determine the appropriate dose of DZ-002; and
* To assess the safety and efficacy of DZ-002.

Participants will receive one of three different doses of the study drug through an IV over a 4-hour period on Days 1, 8, 15, and 22 of a 4-week period, or cycle. During the study, participants will have regular visits to the study clinic and multiple tests for safety and research purposes, including blood tests, along with other tests and scans. Participants will receive the study drug weekly in 4-week (28-day cycles) until there are side effects that cannot be tolerated, there is disease-worsening, or the researchers decide to stop. A post-treatment visit and a 30-day post-treatment follow up visit will be conducted after the last dose of study drug.

Risks of DZ-002 include nausea, vomiting, diarrhea, chills, low levels of red blood cells, low levels of platelets, fatigue, skin rash, low blood pressure, and feeling unwell.

DETAILED DESCRIPTION:
This is an open label, non-randomized, Phase 2 study to asses the efficacy, safety, PK and pharmacodynamic study of DZ-002 in patients with metastatic pancreatic adenocarcinoma who have completed four or more months of first line chemotherapy with a response of stable disease, partial response, or complete response as documented by CT.

There are two parts in this study, a dose escalation part and a dose expansion part. In the dose escalation part of this study, participants will receive one of three different doses of the study drug DZ-002: 5 mg/kg, 6 mg/kg, or 7 mg/kg. Participants will receive the study drug intravenously (into a vein) over a 4-hour period on Days 1, 8, 15, and 22 of a 4-week period. This 4-week period (28 days) is referred to as a cycle.

The first 3 to 6 participants taking part in this study will get the lowest dose of 5 mg/kg. If the drug does not cause worrisome side effects, the next group of 3 to 6 participants in the study will get a higher dose of 6 mg/kg. If the drug does not cause worrisome side effects, the last group of 3 to 6 participants will receive the highest dose of 7 mg/kg. The investigator will watch each group carefully as they increase the dose. The dose will increase for each group until participants have worrisome side effects that require the dose to be lower. Once the highest dose with manageable side effects is found, the dose escalation is stopped.

In the dose expansion part of this study, the highest dose with manageable side effects will be given to 30 more participants. This will help the investigators better understand the side effects that may happen with this drug.

Participation in this study is divided into different visits:

1. Screening Visits
2. Treatment Visits
3. End of Treatment Visits
4. Post-Treatment Visits

Various tests are run during each of these different visits as described below:

* Collection of medical history and current medications
* Physical exam, height, weight, vital signs
* Lung function tests
* CT scans or PET scans
* Heart function tests, such as Echocardiogram or multiple-gated acquisition
* Electrocardiograms (ECG)
* Blood draws for routine lab tests
* Additional blood samples to measure the amount of study drug in blood
* Urine collection
* X-ray, if indicated
* Tumor biopsy, optional
* Pregnancy test, if applicable

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed diagnosis of metastatic pancreatic adenocarcinoma who completed 4 months or more of first line chemotherapy and have achieved at least SD documented by CT scan.
2. Male or female patients ≥18 years of age;
3. Measurable or evaluable disease by RECIST v 1.1;
4. Capable of understanding and complying with protocol requirements;
5. A life expectancy of greater than 8 weeks at Screening;
6. ECOG PS of 0 to 1;
7. Written informed consent from the patient or the patient's legally acceptable representative prior to the initiation of any study procedures;
8. Adequate bone marrow, liver, and renal function as defined below:

   1. Hemoglobin ≥ 10.0 g/dL (transfusions and/or erythropoietic stimulating growth factors allowed);
   2. Absolute neutrophil count ≥ 1500/μL;
   3. Platelet count ≥ 75,000/ μL;
   4. Alanine aminotransferase and aspartate aminotransferase ≤ 2.5 × the upper limit of normal (ULN) or ≤ 5 × ULN for patients with known hepatic metastases;
   5. Total serum bilirubin ≤ 1.5× ULN or ≤ 2 .0 × ULN if liver metastases are present. Patients with a known history of Gilbert's syndrome (≤ 3.0 × ULN)
   6. Estimated creatinine clearance ≥ 40 mL/min (using the Cockcroft Gault formula);
9. Adequate cardiac function as estimated by left ventricular ejection fraction (LVEF) > 50% by multiple-gated acquisition (MUGA) or echocardiogram (ECHO);
10. Adequate pulmonary function tests with FEV 1 >90% and Vital capacity >90%

Exclusion Criteria:

1. New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, a history of risk factors for Torsades de Points, including heart failure, hypokalemia, and family history of long QTc syndrome, or evidence of ischemia on ECG;
2. Baseline QTc exceeding 470 msec (using the Fridericia's formula) and/or patients receiving Class 1A or Class III antiarrhythmic agents or concomitant medications that prolong the QT/QTc interval;
3. Patients with individual pulmonary metastases > 5 cm diameter or with high metastatic burden to the lungs as determined by the principal or the primary investigator;
4. Patients with extensive bone metastases as determined by the principal or the primary investigator;
5. Patients with a current positive COVID-19 diagnosis, or are currently symptomatic with COVID-19, or who have had COVID-19 in the last month, or with a history of COVID-19 diagnosis with respiratory complications;
6. Active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy;
7. Treatment with simvastatin unless it can be stopped prior to and during the study;
8. Treatment with strong inhibitors and inducers of CYP3A4 or narrow therapeutic index substrates of CY3A4, CYP2B6, CYP1A2, CYP2C9, and CYP2C8, unless these can be stopped prior to and during the study;
9. Known sensitivity to DZ-002 or its excipients;
10. Pregnant (confirmed by serum or urine pregnancy test) or is breast feeding;
11. Unwillingness or inability to comply with procedures required in this protocol;
12. Known infection with human immunodeficiency virus and CD4 lymphocyte count ≤ 200 cells/mm3, active hepatitis B virus, or hepatitis C virus infections;
13. Serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor;
14. Patients who are currently receiving any other investigational agent
15. Patients with G6PD deficiency or hereditary methemoglobinemia
16. Patients taking the following medications: Nitroglycerine, dapsone or antimalarials (e.g. chloroquine, primaquine)
17. Patients with known pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Up to 28 days of last patient dosed during the escalation phase
  To determine the RP2D
Incidence of Dose Limiting Toxicities (DLTs) | Up to 28 days
  Dose limiting toxicities refer to toxicities experienced during the first 28 days of DZ-002 treatment that have been judged to be clinically significant and related to study treatment.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Approximately 2 years
  Incidence and severity of treatment-emergent adverse events (TEAEs), as assessed by CTCAE, V5.0.
Progression-Free Survival | Until disease progression (up to 6 months)
  Progression-free survival is defined as the interval from first dose date of study drug (DZ-002) to the earlier of the first documentation of definitive disease progression or death from any cause; definitive disease progression is progression based on RECIST criteria v1.1.
Objective Response Rate (ORR) | Approximately 1 year
  Dose Expansion portion only. The Proportion of participants who achieve complete response (CR) or partial response (PR), as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Pharmacokinetic (PK) Parameter: Cmax of DZ-002 | Predose and up to 24 hours post dose
  Cmax is defined as the maximum observed concentration of DZ-002
Pharmacokinetic (PK) Parameter: Tmax of DZ-002 | Predose and up to 24 hours post dose
  To determine the time of maximum concentration (Tmax) of DZ-002
Pharmacokinetic (PK) Parameter: AUC of DZ-002 | Predose and up to 24 hours post dose
  To determine the area under the curve at the end of the DZ-002 dosing

OTHER OUTCOMES:
Biomarker | From baseline to 30 days after the last dose, or end of study if clinically indicated
  To evaluate potential biomarkers of response by evaluating changes in blood components, including circulating tumor cells (CTCs) in response to treatment with DZ-002.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Becerra, MD, Principal Investigator — Hoag Memorial Hospital Presbyterian
Locations (1):
- Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No